CLINICAL TRIAL: NCT05528393
Title: Prolactin and FGF21 in Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shen Qu (Other)
Responsible Party: Sponsor-Investigator, Shen Qu, Principle investigator, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: gestational diabetes mellitus
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Hyperprolactinemia Pregnancy
Keywords: Gestational Diabetes Mellitus; Prolactin; Insulin resistance; Fibroblast growth factor 21
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM and Non-GDM
  Interventions: Diagnostic Test: Blood sampling
- Pregnant group and non-pregnant group
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — blood sampling

SUMMARY:
Prolactin (PRL) and PRL receptor (PRLR) signaling has been validated to play an important role in the modulation of glucolipid metabolism. However, the role of serum PRL levels in gestational diabetes mellitus (GDM) remains unclear. The investigators aimed to explore the possible influence of serum PRL within or without normal range on the development of GDM.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 45 years
* completed a 75-g oral glucose tolerance test (OGTT)
* females with pregnancy

Exclusion Criteria:

* severe liver and renal dysfunction, preexisting heart disease, malignancy, or endocrine diseases such as pituitary adenoma and hypogonadism
* mental illness
* genetic disease
* current or previous treatment that might affect PRL and insulin secretion
* diabetes before pregnancy
* loss to follow-up, or withdrawal from the study
* unable to understand and comply with the study protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who met the above criteria were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes mellitus (GDM) | 2019-2023
  GDM is defined as a glucose intolerance resulting in hyperglycaemia of variable severity with onset during pregnancy. It can be diagnosed by the criteria: a fasting plasma glucose (FPG) concentration of O126 mg/dl on two separate occasions or a random blood glucose concentration of O200 mg/dl on two separate occasions.
PRL | 2019-2023
  serum prolactin level

SECONDARY OUTCOMES:
Insulin resistance (IR) | 2019-2023
  It was considered to be IR if HOMA-IR >2.5
HOMA-IR | 2019-2023
  It was calculated as: fasting plasma glucose (FPG) x fasting insulin (FINS)/22.5
OGTT | 2019-2023
  OGTT was performed after an overnight fasting in each patient and blood samples were taken at 0, 30, 60, 120, and 180 min to determine the concentrations of plasma glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China